CLINICAL TRIAL: NCT05693584
Title: The Effect of Using Virtual Reality Glasses on Pain During Fistula Cannulation in Hemodialysis Patients: A Randomized Controlled Study
Brief Title: The Effect of Using Virtual Reality Glasses on Pain During Fistula Cannulation in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Hülya Elmali Simsek, Principle Investigator (Dr), Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: fbu_nurs_elmali_001
Record Dates: First submitted 2022-12-26; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Hemodialysis Patients
Keywords: avf cannulation; hemodialysis; pain; virtual reality
MeSH Terms: conditions — Pain | interventions — Osteogenesis, Distraction

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Pain assessments were made by the service nurses, and virtual reality glasses were applied by the researcher. The data were collected by one researcher and the analysis and evaluations were made by the other researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality glasses (Experimental): Experimental group:Group applying virtual reality glasses
  Interventions: Other: distraction
- Routine practices (No Intervention): No procedure was performed on the patients other than the routine practices of the clinic.

INTERVENTIONS:
Other: distraction — diverting the patient's attention with virtual reality glasses
  Arms: Virtual reality glasses

SUMMARY:
Hemodialysis; It is the process of returning the liquid and solute content of the blood taken from the patient to the patient as a result of rearrangement by means of a membrane and with the help of a machine. A permanent vascular access that can be used for months or years is required for HD treatment to be sufficient for patients with end-stage renal disease to survive and improve their quality of life. For this reason, patients who will be treated for HD need to have an arterio-venous fistula (AVF), graft or catheter to ensure adequate blood flow. CRF patients treated with HD are exposed to 300-320 AVF cannulations per year on average. The size and length of the diameter of the fistula needles, the piercing process created in the skin, the advancement of the needles into the tissue during the procedure, the entry angle of the needles and the entry techniques cause the patients to experience pain during the procedure.

Non-pharmacological methods frequently used in pain control include many applications such as distraction, massage, hot and cold application, aromatherapy.

Distraction, which is one of the non-pharmacological methods, is a method that enables patients to focus their attention on a different point and to control and reduce the symptoms they experience. Methods such as listening to music, taking pictures, watching television, solving puzzles, daydreaming, deep breathing and coughing exercises, sphygmomanometer blowing, active listening, tapping, inflating balloons, distraction cards and using virtual reality glasses are used for this purpose.

With the virtual reality glasses, the individual gets away from the environment with the glasses connected to the device worn on his head and the sounds coming from the headset, concentrates his attention on the image he watches and feels like he is in another world thanks to these five-dimensional glasses. The most basic feature that distinguishes virtual reality glasses from similar applications is that it gives people a real feeling. Virtual reality glasses, which are easy to apply and use, have no side effects, and can be effective in physical, psychological and social recovery, are an initiative that can be preferred in health applications.

In this study, it is aimed to determine the effect of using virtual reality glasses on pain during fistula cannulation applied to hemodialysis patients.

The hypotheses of the research; H₀: The use of virtual reality glasses is not effective in reducing the severity of pain.

H1: The use of virtual reality glasses reduces the severity of pain.

DETAILED DESCRIPTION:
The research was carried out with patients in the hemodialysis unit of a private hospital in Istanbul, between September and November 2022.The study had a pre-test post-test design and was a single-center, parallel-design, randomized controlled experimental study.

Priori Power Analysis was performed to determine the sample size and Cohen's standard effect size reference method was chosen accordingly. Considering 85% power, 0.005 significance level, and 0.8 effect size for the study, the minimum required sample size was calculated as 23 for each group. Since it was thought that there might be data loss, it was decided to include 28 patients in each group and 56 patients in total.

Computer-assisted simple randomization (https://www.randomizer.org/) was used to determine the groups. There wasn't any blocking in this simple randomization. There wasn't any blinding for the patients or the researchers throughout the study. Pain assessments were made by the service nurses, and virtual reality glasses were applied by the researcher. The data were collected by one researcher and the analysis and evaluations were made by the other researcher. Thus, blanking was used during data collection and analysis.

The population of the study consists of patients (n=82) in the hemodialysis unit of a private hospital in Istanbul, and the sample consists of patients who meet the research criteria and agree to participate in the study (n=47).

In data collection; Introductory Information Form and Visual Analog Scale (Visual Comparison Scale) (VAS) were used.

Virtual reality glasses: Bobo VR Z4 brand virtual reality glasses with 5.7 inch 1440x2560 pixel screen resolution and JBL brand wireless headset were used.

In this study, it is planned to analyze the data in SPSS program. Normality tests, mean, standard deviation, minimum, maximum, number-percentage distributions in data analysis; Independent Groups t-test, Mann Whitney U test, One-Way Analysis of Variance, Kruskal-Wallis test will be used. Differences between groups in terms of categorical variables will be examined with the chi-square test. Pearson correlation analysis will be used to examine the relationships between variables, and Cohen-d effect size will be used to determine the effect size.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old,
* Regular hemodialysis,
* A single injection from the AVF was attempted,
* Patients who do not have vision or hearing problems and who agree to participate in the study.

Exclusion Criteria:

* Have taken any analgesic in the last 3 hours,
* Redness in the fistula area, signs of infection,
* Does not speak Turkish, has language problems; illiterate patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (Visual Comparison Scale) (VAS) | immediately after intervention
  One end of the VAS is 10 cm or 100 mm, which indicates that the patient has very good, no pain (0 points), and the other end is very bad, unbearable pain (10/100 points). It is a scale that is evaluated by making

SECONDARY OUTCOMES:
Visual Analog Scale (Visual Comparison Scale) (VAS) | 30 minutes after intervention
  One end of the VAS is 10 cm or 100 mm, which indicates that the patient has very good, no pain (0 points), and the other end is very bad, unbearable pain (10/100 points). It is a scale that is evaluated by making

CONTACTS AND LOCATIONS:
Locations (1):
- Medicana Çamlıca Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No